CLINICAL TRIAL: NCT00509535
Title: Prospective, Randomized, Double Blind Comparative Study on the Use of Two Creams in Xerosis Atopic Probands Biomedical Findings With Vitreoscilla Filiformis
Brief Title: Prospective, Randomized, Double Blind Comparative Study on the Use of Two Creams in Xerosis Atopic Probands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oreal (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-AD-003
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2007-07-31 (Estimated); Status verified 2007-07

CONDITIONS: Atopic Dermatitis
Keywords: Vitreoscilla filiformis extract; SCORAD; pruritus; microflora; TEWL
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: vitreoscilla filiformis cream

SUMMARY:
Atopic dermatitis (AD), a chronic and relapsing inflammatory skin disease, is associated with elevated IgE levels and Th2 responses. It is currently believed that non-pathogenic bacteria modulate intestinal immune responses avoiding the development of allergic diseases. However, effects of oral probiotics on AD could not be reproduced in all studies and direct immuno-modulation of the skin associated immune response by non-pathogenic bacteria has not been investigated so far. We therefore performed a double blind placebo controlled clinical study on the effects of an ointment containing 5% extracts of the non-pathogenic bacteria Vitreoscilla filiformis on AD. Seventy-five AD patients (6-70 years of age) were randomized to receive either Vitreoscilla filiformis ointment 5% or vehicle ointment daily for 30 days. Efficacy evaluations, including the "Score of Atopic Dermatitis" (SCORAD), transepidermal water loss, assessement of microflora, and the patient assessment of itch and loss of sleep occurred at baseline, day 15, and day 29.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronically relapsing inflammatory skin disease and often coexists with other atopic diseases, such as allergic rhinitis, conjunctivitis and asthma (Biedermann and Röcken 1999, Biedermann et al. 2001, 2004, 2006; Leung et al., 2000, 2003a, 2003b). Even though the immune pathology of AD is not precisely understood, today the new concept of atopic dermatitis pathology is based on a large set of data. In most patients with AD, dry skin and dysfunction of the epidermal barrier is found. As an important prove of concept, the loss of function mutation of the epidermal protein filaggrin impairing skin barrier function was found and can be detected in about 15% of kaukasian AD patients (Palmer et al., 2006). As a consequence, patients with AD are predisposed to develop sensitizations dominated by a Th2 immune phenotype (Hudson, 2006).

Independently of the filaggrin study, it was demonstrated earlier that a disrupted barrier function of the stratum corneum is present in atopics not only in involved skin, but also in uninvolved dry skin facilitating permeation of various environmental substances into the skin (Berardesca et al., 1990; Werner et al., 1985; Watanabe et al., 1991; Loden et al, 1992). As a biomarker, an increased level of transepidermal water loss (TEWL) can be demonstrated (Tagami et al., 1985; Ghadially et al., 1996). Various functional and morphological studies on atopic xerosis that clinically appeared without inflammation demonstrated that cellular inflammation is already present in atopic skin and a key and initial step in the development of atopic dermatitis (Watanabe et al., 1991; Uehara et al., 1984). In fact, barrier dysfunction, atopic immune dysregulation, and atopic dermatitis pathogenesis are not independent events, but closely linked (Biedermann 2006; Hudson 2006). Th2 lymphocytes dominate the atopic immune phenotype and are the underlying cell type responsible for the induction if IgE antibodies (Biedermann et al. 1999, 2004). Barrier dysfunction predisposes for the development of Th2 lymphocytes and Th2 cells are the first cell type invading atopic skin initiating inflammation and the inflammatory vicious circle of inflammation (Biedermann 2002; 2004; Lametschwandtner et al. 2004; Günther et al. 2005). Next to Th2 lymphocytes, in atopic dermatitis skin lesions, infiltrates of eosinophils and cells of the mononuclear phagocyte lineage are found.

The altered skin structure of people with atopic predisposition allows increased penetration of allergens and irritative substances (Roll et al., 2004; Hudson 2006). Many studies have shown that the extent of S. aureus colonization correlates with AD disease activity (Cho et al., 2001; Biedermann 2006). In more than 90% of AD patients, a massive skin colonization with S. aureus (up to 107cfu/cm2 of lesional skin) can be found (Matsui et al., 2000). A prerequisite for bacterial colonisation are the genuine barrier dysfunction, mechanical disruption of the barrier and trigger of inflammation (scratching), alkaline pH, decreased IgA secretion through sweat production, predominant Th2 cells inhibiting anti-infectious immune responses, and reduced antimicrobial peptides, all representing important pathophysiological features leading to the disruption of the primary skin defense system (Biedermann et al. 2001; Biedermann&Röcken 2001,; Biedermann et al. 2002; Biedermann 2006; Howell, 2005; Rieg 2005).

Among several microbes colonising the skin, the bacterium Staphylococcus aureus (S. aureus) may play the most important role in the pathogenesis of dermatitis of atopic people (Biedermann 2006). This colonization is observed not only in the involved inflammatory skin but also in the non involved dry skin. The ratio Staphylococcus aureus / Staphylococcus epidermidis is inverse in comparison to healthy skin. Many studies have shown that the extent of S. aureus colonization correlates with AD disease intensity (Cho et al., 2001).

Reduced expression of antimicrobial peptides was demonstrated for AD skin and favours colonization with S. aureus (Ong et al. N. Engl. J. Med. 2002; Howell et al.. Immunity. 2006;24:341-8; Rieg et al. JI 2006). In addition, dry skin may by itself allow colonization with bacteria such as S. aureus. Decreased levels of sphingosine, which has antimicrobial properties and the fact that S. aureus itself stimulates the hydrolysis of ceramides by bacterial derived ceramidase in atopic skin add the dysfunction of the immune barrier in AD (Arikawa et al., 2002; Kita et al, 2002). The cell membrane of S. aureus contains adhesins for epidermal and dermal laminin and fibronectin allowing attachemment of S. aureus. to the skin and these docking positions for S. aureus are uncovered in lesional skin (Cho et al, 2001). The precise mechanism by which S. aureus gains access to the dermis is unknown, but it is suggested that again IL-4, produced by T helper type 2 cells, induces fibronectin synthesis, which in combination with plasma exsudation of fibrinogen, allows S. aureus to bind to the skin. Moreover, S. aureus is able to encase itself in a kind of biofilm composed of a hydrated matrix of polysaccharides (glycocalix) and proteins, which supports cell adhesion (Akiyama et al., 2003). After colonization, S. aureus contributes to skin inflammation e.g. by secreting toxins and an array of so called pathogen associated molecular pattern (PAMP) that bind their pathogen recognition receptors such as Toll- like receptors and directly triggering inflammation (Biedermann 2006). Moreover, S. aureus PAMPs also influence T cell mediated skin inflammation by indirectly regulating skin homing of T cells and orchestrating chronic inflammation in AD skin (Biedermann 2006; Biedermann et al. 2006).

Vitreoscilla filiformis (Vf) (ATCC15551) used in this study is a non-photosynthetic, non-fruiting gliding bacteria as defined according to the classification of Bergey's (1989). This filamentous bacterium belongs to the order of Beggiatoales. It is a micro-organism found in sodic sulphuretted thermal springs recognized for their local anti-pruriginous and anti-inflammatory properties.

The micro-organism Vitreoscilla filiformis (Vf) was cultivated on a defined and sterile medium, expanded and isolated to constitute a biomass called "pure extract of thermal plankton". The term plankton describes the zooplankton (chemiotrope microorganisms) in contrast to the phytoplankton (phototrope microorganisms). At the end of culturing, the biomass is concentrated by stabilized centrifugation and autoclaved.

The technical preparation is a sterile aqueous suspension of the plankton. In vitro studies show that this plankton supports the production of collagen by fibroblasts and reinforces the antioxidants systems; it prevents Langerhans cell alterations (reconstructed skin or organotypic skin culture) exposed to UVB. It exhibits non-specific immunomodulatory effects on cellular immunity and in particular on macrophages (Patent US, 6,190,671 B1; US, 6,242,229 B1; WO-94/02158).

Preclinical studies showed that this extract has anti-inflammatory activities (decreases ear oedema after acid arachidonic treatment and modulates contact hypersensitivity reaction with oxazolone). Moreover, this new compound promotes healing of epidermis and dermis (scaring following suction blister or following incision in preclinical studies; Patent US, 6,190,671 B1). Therefore, this new compound promises to alleviate infections usually found on the skin after skin burning, protects skin against ultraviolet alterations and displayss moisturizing properties for the skin.

Clinical trials showed that the bacterial extract Vitreoscilla filiformis is effective against acne and seborrhoeic dermatitis and promotes moisturization of the skin (studies in Seoul, Korea and in Nice, France and patent FR-2,283, 223) and has been shown to be beneficial for sensitive skin (clinical trial by Dr Desruelle F in Nice, France) Moreover, a randomized, double-blind, placebo-controlled trial with a formulated 5% extract of Vitreoscilla filiformis on symmetric active lesions of AD according to a split-body design was performed with Prof. J. F. Nicolas in Lyon, France.

In this study, the treatment (applied twice daily) with the cream containing 5% Vitreoscilla filiformis extract was found to be safe and well tolerated. Moreover, this extract significantly alleviated AD in older children (from 7 years old) and adults compared with vehicle treatment (p=0.008; Wilcoxon signed ranks test). The therapeutic effects of the extract were observed within the second week of the application and steadily increased thereafter. This effect of the cream containing 5% Vitreoscilla filiformis extract appeared to have a rapid onset especially in regard to pruritus as demonstrated using the mEASI index. Paired testing confirmed a significant difference in the decrease of pruritus on the 5% Vitreoscilla filiformis extract treated side at day 28 (p=0,046, Wilcoxon exact signed ranks test). (Gueniche et al. 2006).

Our task was to perform a double blind randomized prospective study comparing 5% Vitreoscilla filiformis extract (cream B) whith its vehicle (cream A) including measurements of biometric changes occurring during the use of the two creams.

During the study biometrical and clinical measurements including the transepidermal water loss, the qualification and quantification of skin microflora and the clinical evaluation of the skin findings before, during and after the use of the creams was documented. Further the proband's experiences with the use of the creams were assessed. Biometric variables of the skin are determined before, during and after the use of cream A and cream B.

The transepidermal water loss as biometrical value was estimated to assess the skin barrier function at all visits.

We evaluated if topical application of cream A and cream B influenced the microflora of skin of atopic volunteers. Qualification and quantification of several bacteria (S. aureus, S. epidermis, P. acnes, Streptococci, E. coli) was performed before, during and at the end of the study period.

In addition, the intensity of pruritus and the clinical aspect of the skin was assessed.

At the end of the study each volunteer filled out a questionnaire asking about oiliness, distribution, consistency and adsorption of the creams.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild atopic dermatitis are included.
* The eczematous lesions may not pass over 5% of the total body surface.
* The lesions may not weep.

Exclusion Criteria:

* Past history of severe scaring by skin surgery
* Past history of cutaneous cancer, malignant melanoma
* Patient who show a lack of compliance
* Currently participating or having participated in another clinical trial during the last 3 months prior to the beginning of this study
* Allergy or incompatibility of one of the components of the cream
* Pregnant or breast feading woman
* Retraction of the written informed consent

  * Patients who cannot keep untreated with topical steroids are not included. Patients with severe or infected atopic dermatitis are excluded
  * patients where conventional antiinflammatory therapy cannot be withdrawn are excluded

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2005-01; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation SCORAD. In addition a visual analogue scale for subjective estimation of pruritus | at day 0 (visit 1), at day 15 (visit 2) and at least at day 29 (visit 3).

SECONDARY OUTCOMES:
• Evaluation of TEWL • Qualitative and quantitative analyses of skin microflora • Proband's questionnaire about oiliness, distribution, consistency and adsorption of the creams | day 0 (visit 1), at day 15 (visit 2) and at least at day 29 (visit 3).

CONTACTS AND LOCATIONS:
Overall Officials: Tilo Biedermann, Pr PhD, MD, Principal Investigator — Eberhard Karls University
Locations (1):
- Eberhard karls University-Dept Dermatology, Tübingen, Germany